CLINICAL TRIAL: NCT05611411
Title: The Exploration of Maximum Alveolar Concentration of Sevoflurane for Maintaining Effective Spontaneous Respiration
Brief Title: Maximum Alveolar Concentration of Sevoflurane for Maintaining Effective Spontaneous Respiration
Acronym: MaACesr
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, Chief anesthesiologist, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2022ZSLYEC-493
Record Dates: First submitted 2022-11-06; First posted 2022-11-10 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Sevoflurane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation will bring many adverse effects. Positive pressure can affect hemodynamics. Inhalation of higher concentrations of oxygen during mechanical ventilation can result in reabsorbed atelectasis for the lungs with a low ventilation-perfusion ratio. Patients who are intubated and mechanically ventilated are at risk for ventilator-associated pneumonia. Mechanical ventilation can induce or aggravate lung injury, called ventilator-induced lung injury (VILI) , Minimizing the duration of mechanical ventilation is the best way to reduce complications.

Sevoflurane is a halogen group of inhaled anesthetics commonly used in clinical, with sedation, analgesia, muscle relaxation. Sevoflurane also inhibited respiratory function, tidal volume decreased with the depth of anesthesia, respiratory rate increased, higher than the conscious respiratory rate, but not enough to fully compensate for the decreased tidal volume. The results showed that with the increase of the depth of anesthesia, the minute ventilation decreased, and the ability to remove carbon dioxide also decreased.

Based on the background of the study and the pharmacological properties of sevoflurane, we sought to explore the maximum alveolar concentration of sevoflurane for maintaining effective spontaneous respiration in patients, i.e.FiO2 = 30% , PaO2 > 92% , VT > 5 ml/kg, RR > 8/min, PETCO2 < 50 mmHg, sustained > 20s, the time from the beginning of inhalation induction to 1 point OAAS, the changes of hemodynamics during induction, and the recall of induction and operation were also explored.

DETAILED DESCRIPTION:
Mechanical ventilation is the most widely used short-term life support technique in the world, which can not only provide good condition for anesthesiologists to manage airway, it can also prevent respiratory muscle fatigue and carbon dioxide accumulation caused by insufficient ventilation.

At the same time, mechanical ventilation will also bring a lot of adverse effects. Positive pressure ventilation can affect hemodynamics, and studies have shown that high intrathoracic pressure, especially high plateau pressure, can adversely affect right ventricular afterload and function. Inhalation of higher concentrations of oxygen during mechanical ventilation can result in reabsorbed atelectasis for the lungs with a low ventilation-perfusion ratio. Patients who are intubated and mechanically ventilated are at risk for ventilator-associated pneumonia due to low oral and pharyngeal secretions, reduced cough efficiency, and impaired mucociliary clearance. Mechanical ventilation can induce or aggravate lung injury, called ventilator-induced lung injury (VILI) .

Minimizing the duration of mechanical ventilation is the best way to reduce complications.

Sevoflurane is a halogen group of inhaled anesthetics commonly used in clinical, with sedation, analgesia, muscle relaxation. The blood/gas distribution coefficient is low and the effect is quick. The elimination mainly depends on the lung exhalation, about 5% passes through the liver metabolism, is affected by the anaesthesia time long little. Long-term low-flow sevoflurane inhalation anesthesia has little effect on liver and kidney function.

Sevoflurane also inhibited respiratory function, tidal volume decreased with the depth of anesthesia, respiratory rate increased, higher than the conscious respiratory rate, but not enough to fully compensate for the decreased tidal volume. The results showed that with the increase of the depth of anesthesia, the minute ventilation decreased, and the ability to remove carbon dioxide also decreased.

Based on the background of the study and the pharmacological properties of sevoflurane, we sought to explore the best alveolar concentration of sevoflurane for maintaining effective spontaneous respiration in patients, i.e. FiO2 = 30% , PaO2 > 92% , VT > 5 ml/kg, RR > 8/min, PETCO2< 50 mmHg, sustained > 20s, the time from the beginning of inhalation induction to 1 point OAAS, the changes of hemodynamics during induction, and the recall of induction and operation were also explored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-60 years old
2. ASA gradeⅠ~Ⅱ
3. Scheduled for elective surgery under general anesthesia with tracheal intubation

Exclusion Criteria:

1. Elective head and neck and chest surgery patients;
2. Chronic respiratory disease or acute respiratory infection;
3. Indication of difficult airway during preoperative visit;
4. Risk of reflux aspiration;
5. Did not receive regular antihypertensive therapy or blood pressure was not well controlled；
6. Severe organic heart disease;
7. Abnormal function of liver and kidney;
8. Allergic to inhaled anesthetics and known or suspected genetic history of malignant hyperthermia;
9. Mental disorders or long-term history of taking psychotropic drugs and cognitive impairment;
10. History of drug abuse and alcohol abuse;
11. Pregnant or nursing;
12. Participated in any clinical trial as a subject within the last 3 months;
13. Refuse to participate or do not sign or refuse to sign an informed consent form;

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for elective surgery under general anesthesia with tracheal intubation，with better general situation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-03 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
MaACesr | 2022.12.01-2023.06.01
  maximum alveolar concentration of sevoflurane for maintaining effective spontaneous respiration

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China